CLINICAL TRIAL: NCT02134990
Title: A Phase IIa, Open-Label, Single- Center Study to Assess the Activity of Oshadi D and Oshadi R in Combination With Docetaxel, as 2nd Line Therapy for Metastatic Non Small Cell Lung Cancer
Brief Title: Oshadi D and Oshadi R in Combination With Docetaxel, as 2nd Line Therapy for Metastatic Non Small Cell Lung Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Oshadi Drug Administration (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OS-LC-P2a-01
Record Dates: First submitted 2014-05-07; First posted 2014-05-09 (Estimated); Last update posted 2018-04-18 (Actual); Status verified 2018-04

CONDITIONS: Carcinoma, Non-Small-Cell Lung
Keywords: Carcinoma, Non-Small-Cell Lung; Docetaxel
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Docetaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Oshadi D and Oshadi R with Docetaxel (Experimental): Oshadi D and Oshadi R anti cancer agents with Docetaxol chemotherapy
  Interventions: Drug: Oshadi D and Oshadi R; Drug: Docetaxel

INTERVENTIONS:
Drug: Oshadi D and Oshadi R — Anti cancer agents
Drug: Docetaxel — Chemotheraphy
  Other Names: Taxoter

SUMMARY:
The study will be a prospective open-label single-center study in previously treated patients with Non Small Cell Lung Cancer (NSCLC). Treatment efficacy and safety of the combination of Oshadi D and Oshadi R with Docetaxel will be will be evaluated.

Patients will receive Docetaxel in combination with Oshadi D and Oshadi R. Patient will be evaluated throughout the study for safety and tolerance to multiple dose regimens of Oshadi D and Oshadi R.

CT or MRI imaging will be performed prior to treatment initiation and at the end of every 3 Docetaxel cycles (12 weeks). In case of disease progression, dose augmentation will be considered or subsequent therapy.

ELIGIBILITY:
Inclusion Criteria:

* Locally advanced or metastatic NSCLC (IIIB-IV)
* Failure of first line anti-cancer therapy (either radiological documentation of disease progression or due to toxicity) in advanced disease or subsequent relapse of disease following first line therapy
* Man or woman 21 years and above
* Adequate performance status (ECOG 0, and 1)
* Patient must have adequate organ function
* Written informed consent
* Females of childbearing potential and males must be willing to use an effective method of contraception (hormonal or barrier method of birth control; abstinence) from the time consent is signed until 6 weeks after treatment discontinuation.
* Females of childbearing potential must have a negative pregnancy test within 7 days prior to being registered for protocol therapy.

Exclusion Criteria:

* Any treatment with investigational agent within 10 days prior to registration for protocol therapy.
* Cerebrovascular accident, transient ischemic attack or myocardial infarction within 3 months prior to registration for protocol therapy.
* Evidence of pulmonary embolism within 3 months prior to registration for protocol therapy.
* Any history of hematologic malignancies.
* Patient with known positive HIV serology at screening.
* Female patient who are breastfeeding or have a positive pregnancy test at screening or at any time during the study.
* Uncontrolled hypertension (>160/100 mm Hg despite optimal medical therapy).
* Evidence of ongoing cardiac dysrhythmias of NCI CTCAE (Common Toxicity Criteria for Adverse Effects) Version 3.0 grade 2.
* Patients in whom radiation or surgery is indicated
* Significant swallowing disorders.
* Small bowel surgery.
* Suspicion of absorption disruption as a result of abdominal radiation
* Pre-existing mal absorption syndrome, irritable bowel syndrome or other clinical situation which could affect oral absorption.
* Evidence of concurrent (< 5 years) second malignancy
* Mental disorders.
* Inability to give written informed consent.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2014-06 (Actual); Primary Completion 2019-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
overall survival time | 12 months
  overall survival of the patient

SECONDARY OUTCOMES:
Adverse events and serious adverse events occurence | One month following treatment initiation
  Adverse events and serious adverse events occurred during the study
Patient report outcome | 12 months
  To assess patients quality of life by QLC30 questionnaire

OTHER OUTCOMES:
Progression Free Survival (PFS) | 12 months
  time from treatment initiation to documentation of disease progression or death)
Duration of Response (DoR); | 12 months
  response duration to the drug
Change in tumor size | 12 weeks
  changes in tumor size

CONTACTS AND LOCATIONS:
Overall Officials: Hovav Nehushtan, Prof., Principal Investigator — Hadassah Medical Organization
Locations (1):
- Hadassah Medical Center, Jerusalem, Israel